CLINICAL TRIAL: NCT01952431
Title: Measurement and Evaluation of Total Lung Capacity (TLC) in the Field of Pulmonary Functional Testing (PFT)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: PulmOne Advanced Medical Devices, Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: PulmOne-1.0
Record Dates: First submitted 2013-06-13; First posted 2013-09-30 (Estimated); Last update posted 2014-11-11 (Estimated); Status verified 2013-09

CONDITIONS: TLC in Patients With and Without Respiratory System Disease
Keywords: Total Lung Capacity
MeSH Terms: interventions — Total Lung Capacity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PulmOne MiniBox PFT (Experimental): Total Lung Capacity (TLC) testing with PulmOne MiniBoxPFT
  Interventions: Device: Total Lung Capacity (TLC) testing
- ZAN500 (Active Comparator): Total Lung Capacity (TLC) testing with ZAN500.
  Interventions: Device: Total Lung Capacity (TLC) testing

INTERVENTIONS:
Device: Total Lung Capacity (TLC) testing — Comparison of TLC results
  Other Names: TLC

SUMMARY:
A comparative study to test the efficacy of a novel device - the MiniBoxPFT, in measuring TLC (total lung capacity) compared to TLC measured by standard body plethysmography using the ZAN 500. The study will be conducted as a prospective two-arm, open, randomized comparative study.

DETAILED DESCRIPTION:
This study is a prospective, multi-centered, randomized, comparative study designed to demonstrate substantially equivalence performance of the proposed device, the PulmOne MiniBoxPFT, to its predicate device, the ZAN500, for the measurement of total lung capacity (TLC).

ELIGIBILITY:
Inclusion Criteria:

1. Subject is at least 18 years of age.
2. Subject is cooperative and capable of following instructions.
3. Healthy subjects:

   1. Never smokers.
   2. No known history of respiratory, cardiovascular, hepatic, renal or metabolic disease.
   3. BMI < 35.
   4. No persisting respiratory symptoms during the last 12 months. (e.g., dyspnea, chronic cough, wheezing or phlegm).
   5. No history suggesting upper respiratory infection during the three weeks prior to testing.
4. Patients with known disease affecting the respiratory system, with previous documentation of obstructive, restrictive, or mixed obstructive plus restrictive ventilatory abnormality.

Exclusion Criteria:

1. Subjects who are unable to satisfactorily perform routine, full lung function testing(due to non-compliance or claustrophobia).
2. Subjects unable or unwilling to give informed consent.
3. Subjects who have performed any significant physical activity during 1 hour prior to the Study.
4. Patients with a tracheostomy.
5. Pregnant women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2013-04; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Total Lung Capacity (TCL) | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Mordechai Yigla, MD, Principal Investigator — Rambam University Medical Center
Locations (1):
- Rambam University Medical Center, Haifa, Israel